CLINICAL TRIAL: NCT04238442
Title: Assessing the Accuracy of the A&D TM-2657W Oscillometric Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: A&D Medical (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00079695
Record Dates: First submitted 2019-10-01; First posted 2020-01-23 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BP oscillometric measurement (Experimental): Oscillometric BP measurement
  Interventions: Device: A&D TM-2657W oscillometric device

INTERVENTIONS:
Device: A&D TM-2657W oscillometric device — Assessing the accuracy of the A&D TM-2657W oscillometric device using International Standards Organization validation protocol. This involves comparing the accuracy of the A&D device to 2 observer mercury auscultation (gold standard).

SUMMARY:
The A&D automatic blood pressure device is a new kiosk that can measure blood pressure in the general population.

The investigators plan to use the existing International Standards Organization validation protocol to determine whether this device measures blood pressure accurately.

DETAILED DESCRIPTION:
Methods and Analysis

Study methodology will follow the ISO protocol:

* 85 adult (age 18 years or greater) subjects will be included (it is estimated that approximately 140 subjects will need to be screened as some will be ineligible). 85 is the recommended sample size for validation studies using the ISO protocol.
* Subjects will be recruited via an existing registry of over 250 individuals that have participated in past measurement studies, through advertisements, and from the University of Alberta Hypertension Clinic.
* Specific requirements for a certain percentage of subjects with specific age, sex, upper arm circumference, and baseline blood pressure levels will be observed to ensure that a representative sample is studied (according to the ISO standards).
* Subjects that are pregnant or with atrial fibrillation will be excluded. Blood pressure measurements will be taken using recommended, optimal technique.
* Nine measurements will be taken in each subject, alternating between blinded two-observer auscultation with a mercury-based sphygmomanometer (the reference standard) and the TM-2657. Careful attention will be paid to ensuring proper cuffing. The first two measurements will be discarded and the latter seven measurements (4 auscultatory and TM-2657 measurements) will be used in the analysis, which will be conducted according to ISO standards.
* Accuracy will be assessed according to Criterion 1 and 2 of the ISO standard. Bland-Altman plots will be generated. A plot of measurement error versus arm circumference will be generated as well.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* normal sinus rhythm
* have capacity to give consent
* following the International Standards Organization criteria for: gender distribution, limb size, blood pressure distribution

Exclusion Criteria:

* atrial fibrillation
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Accuracy per International Standards Organization Protocol | 3 months
  Agreement of the device to mercury auscultation.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ringrose, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No